CLINICAL TRIAL: NCT04830618
Title: Aberrant DNA Methylation Maker for Predicting Metachronous Recurrence After Endoscopic Resection of Gastric Neoplasms
Brief Title: Aberrant DNA Methylation to Predict Metachronous Gastric Neoplasms
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Dong Ho Lee, M.D., Ph.D., Seoul National University Hospital
Other Study IDs: B-1204/152-004
Record Dates: First submitted 2021-03-31; First posted 2021-04-05 (Actual); Last update posted 2021-04-05 (Actual); Status verified 2021-03

CONDITIONS: Metachronous Neoplasm; Gastric Cancer; Gastric Neoplasm; Aberrant DNA Methylation
MeSH Terms: conditions — Neoplasms, Second Primary; Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study is a prospective cohort study to investigate whether aberrant DNA methylation can be useful for the prediction of metachronous recurrence after endoscopic resection of gastric neoplasms (dysplasia or cancer). From 2012 to 2017, 300 patients were prospectively enrolled after endoscopic resection (ER) of gastric dysplasia or early gastric cancer. All lesions were assessed by endoscopy and biopsy before ER. Endoscopic mucosal resection (EMR) or endoscopic submucosal dissection (ESD) was performed for gastric dysplasia and early gastric cancers which met the absolute indication (differentiated adenocarcinoma, intramucosal cancer, lesions < 20 mm, and no endoscopic evidence of ulceration). All lesions were curatively resected; if non-curatively resected, the patients were not enrolled from the study. All subjects, who provided informed consent, were asked to complete a questionnaire under the supervision of a well-trained interviewer. The questionnaire included questions regarding demographic data (age, sex), socioeconomic data (smoking, alcohol, and education), their family history of GC in first-degree relatives, and history of H. pylori eradication therapy. Also, MOS methylation level at baseline was measured from noncancerous gastric mucosae at corpus. When H. pylori was positive by CLOtest or histology at baseline or during the follow-up, eradication therapy was done. To evaluate whether H. pylori was eradicated, 13C-urea breath testing was performed at least 4 weeks after completion of the eradication therapy. All study subjects were closely followed up since recurrent tumors at previous endoscopic resection sites can be easily detected on endoscopy with biopsy and treated during follow-up. Patients with local recurrence underwent further treatments, including repeated ESD, APC, and gastrectomy based on pathology, and patients who refused treatment received supportive care. All patients underwent endoscopy with biopsy within 6 months, then at 12 months after ESD to check for metachronous lesions or local recurrences. After 12 months, endoscopy with biopsy was performed annually. In case of EGCs, abdominal CT scan was performed in the first year and biennially thereafter to detect lymph node or distant metastases. The definition of the completion of the study protocol was 1) endoscopic and/or radiologic follow-up for more than 3 years, or 2) development of metachronous gastric neoplasm (primary outcome: gastric dysplasia or cancer) during the follow-up. Metachronous recurrence was defined as secondary dysplasia or cancers detected > 1 year after initial diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent endoscopic resection of gastric neoplasms (dysplasia or early gastric cancer)
* All gastric neoplasms at diagnosis should be curatively resected before enrollment.

Exclusion Criteria:

* Previous history of all cancers.
* Previous history of gastrectomy
* Non-curative resection of gastric neoplasms
* Refusal to consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with gastric neoplasms (gastric dysplasia or early gastric cancer) which was curatively resected endoscopically.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2012-09-11 (Actual); Primary Completion 2017-11-16 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Metachronous recurrence | at least > 1 year after enrollment (initial diagnosis), from enrollment to Dec 2020
  Metachronous recurrence was defined as secondary dysplasia or cancers detected > 1 year after initial diagnosis.

REFERENCES:
- [Derived] Shin CM, Kim N, Yoon H, Choi YJ, Park JH, Park YS, Lee DH. Aberrant DNA Methylation Maker for Predicting Metachronous Recurrence After Endoscopic Resection of Gastric Neoplasms. Cancer Res Treat. 2022 Oct;54(4):1157-1166. doi: 10.4143/crt.2021.997. Epub 2022 Jan 18. PMID 35038821